CLINICAL TRIAL: NCT02540070
Title: Ultrasound Guided Motor Sparing Knee Blocks With or Without Dexmedetomidine for Postoperative Analgesia Following Knee Arthroplasty: a Randomized Double Blinded Study
Brief Title: Evaluation of Motor Sparing Knee Block to Infiltration Analgesia for Pain Following Knee Arthroplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104373
Record Dates: First submitted 2014-03-17; First posted 2015-09-03 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis; Knee Arthroplasty; Pain Management
Keywords: Adductor canal Block; ultrasound; periarticular injections; Dexmedetomidine
MeSH Terms: conditions — Osteoarthritis; Agnosia | interventions — Ropivacaine; Epinephrine; Morphine; Ketorolac; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Periarticular (Active Comparator): Patients in group 1 will receive periarticular infiltration of LA mixture (100 ml) consisting of 0.3% ropivacaine, 2.5 µg/mL of epinephrine, 10 mg of morphine and 30 mg of ketorolac at the end of surgery and sham injections of saline into the motor sparing knee blocks preoperatively.
  Interventions: Procedure: Periarticular; Drug: Ropivacaine; Drug: epinephrine; Drug: morphine; Drug: Ketorolac; Drug: saline
- Motor free (Experimental): Patients in group 2 will receive motor sparing knee blocks with 0.5% ropivacaine with 2.5 µg/mL of epinephrine, 30 mg of ketorolac and 10 mg of morphine with a total local anesthetic volume of 60 ml (300 mg). Sham injections of saline (100 ml) will be injected periarticularly at the end of surgery.
  Interventions: Procedure: Motor free; Drug: Ropivacaine; Drug: epinephrine; Drug: morphine; Drug: Ketorolac; Drug: saline
- Motor free with Dex (Experimental): Patients in group 3 will receive motor sparing knee blocks with 0.5% ropivacaine with 1 µg/Kg of dexmedetomidine, 30 mg of ketorolac and 10 mg of morphine with a total local anesthetic volume of 60 ml (300 mg). Patients in group 3 will receive sham injections of saline (100 ml) periarticularly at the end of surgery.
  Interventions: Procedure: Motor free with dex; Drug: Ropivacaine; Drug: morphine; Drug: Ketorolac; Drug: Dexmedetomidine; Drug: saline

INTERVENTIONS:
Procedure: Periarticular
  Arms: Periarticular
Procedure: Motor free
  Arms: Motor free
Procedure: Motor free with dex
  Arms: Motor free with Dex
Drug: Ropivacaine
Drug: epinephrine
  Arms: Motor free; Periarticular
Drug: morphine
Drug: Ketorolac
Drug: Dexmedetomidine
  Arms: Motor free with Dex
Drug: saline

SUMMARY:
Patients undergoing primary total knee replacement will receive either motor sparing knee block to be performed by anesthesia or periarticular local anesthetic infiltration at the end of surgery by surgeons to assess pain relief as well as capacity to ambulate early. The motor sparing knee block will be performed prior to surgery using ultrasonography and the effect of adding dexmedetomidine, an alpha 2 agonist to the injectate with regards to prolonging the duration of analgesia will be assessed.

DETAILED DESCRIPTION:
This prospective randomised double blind study will be conducted on 90 patients undergoing primary total knee arthroplasties of American society of anesthesiologists physical status (ASA) 1-3 class. Patients will be educated regarding verbal rating score (0=no pain; 10= worst pain ever) and postoperative rehabilitation exercises by the physiotherapy. Preoperative motor power will be recorded by a physiotherapist in all patients. All patients will receive pre-operative multimodal analgesia with Tylenol, Naproxen, gabapentin and granisetron which will be continued for at least 5 postoperative days. Patients will be grouped according to the study arm as group 1 (periarticular infiltration of 100 ml of 0.3% ropivacaine with 30 mg of ketorolac, 10 mg morphine and 2.5µg/ml of epinephrine), group 2 (60 ml of 0.5% ropivacaine with 30 mg of ketorolac, 10 mg morphine and 2.5µg/ml of epinephrine) or group 3 (60 ml of 0.5% ropivacaine with 30 mg of ketorolac, 10 mg morphine and 1µg/Kg of dexmedetomidine).

Pre-procedural scan will identify suitable location to perform the three injections. The continuous adductor canal block will be performed under ultrasound guidance in the supine position with the leg in external rotation. The femoral artery is traced from the groin region under the Sartorius muscle until the superior geniculate artery is seen to take off from the femoral artery. This will mark the site of final catheter tip location. The probe will be rotated 900 and moved cephalad tracing the Sartorius and the femoral artery in the long axis till 8cms proximally which will be marked as the needle entry point. The intermediate cutaneous nerve of thigh usually travels as a dual nerve between the Sartorius and rectus femoris above the fascia lata which is identified at this point. Following sterile precautions, the skin will be anesthetized with 1% lidocaine and an 8 cm block needle will be inserted out of plane with the artery in short axis under the Sartorius. The needle will be initially directed laterally to lie above the fascia lata between the Sartorius and rectus femoris muscle and 5 ml of study drug will be injected while withdrawing the needle. The needle is then redirected to enter the fascia of the Sartorius to deliver an additional 5ml of the study drug. The needle is then advanced till the needle tip is seen to lie adjacent to the femoral artery under the Sartorius. Following this, the US probe is rotated to see the Sartorius in the long axis with the artery in the long axis underneath it. The needle is advanced hydrodissecting with 0.5% dextrose until the needle tip is positioned just proximal to the origin of the superior geniculate artery. A block catheter will be inserted 3cms beyond the tip of the needle under US guidance. Following this, 15 ml of test drug will be injected watching for confirmation of STUDY DRUG deposition around the artery. The final catheter tip location will be confirmed with color Doppler as well as pulse wave Doppler and is deemed adequately positioned if seen close to the artery. Following adductor canal block, sartorius will be traced to its origin at the anterior superior iliac spine and lateral cutaneous nerve of thigh will be blocked in the lacuna musculorum between the origin of Sartorius and tensor fascia lata muscle with 10 ml of the study drug. Following the anterior injections, an 8 cms block needle will be inserted near the medial femoral epicondyle under ultrasound guidance and 25 ml of test drug will be injected from the medial epicondyle to the lateral epicondyle between the bone and popliteal artery which constitutes posterior pericapsular injection. Hence, a total volume of 60 ml will be used.

All patients will be enrolled on an intention to treat analysis basis and the block characteristics will be documented on all the aspects of the knee joint by a blinded observer comparing it to the opposite side. Motor power will be tested with a hand held dynamometer before and 20 minutes after the performance of the blocks. Proprioception and vibration will be tested and documented by the same observer before and 20 minutes after the blocks. All patients will receive spinal anesthesia with 15 mg of hyperbaric bupivacaine for the surgery with titrated sedation intraoperatively to a Ramsay sedation score of 3 with propofol 9mg/ml and 1mg/ml of ketamine. The patients will be assessed for pain during rest and activity immediately after the effects of spinal anesthetic wears off (Bromage score of 1), every 2 hourly for 6 hours and at 6, 12 , 24, 36 and 48 AND 72 HOURS. All patients will be evaluated for their readiness to perform physiotherapy after full recovery FROM SPINAL ANESTHESIA (Bromage score of 1), lack of postural hypotension AS ASSESSED BY THE CAREGIVER AND THE PHYSIOTHERAPIST. The adductor canal catheter will be bolused with 10 ml of 0.2% ropivacaine once the patient reports >6/10 anterior knee pain and an infusion will be started at a basal rate of 6ml/Hr with patient controlled boluses (PCRA) of 4ml every 30 minutes as needed. Second rescue analgesia consists of oxycodone 5-10mg every 3-4 hourly. The predominant site of pain will be documented. All patients will be assessed for performance of "Timed up and Go" test at 6 postoperative hours and at discharge. Patients will be deemed to attain discharge readiness if pain and nausea are controlled on oral medications, absence of medical or surgical complications and are able to do five steps in the physiotherapy department. The number of patients that achieved the discharge criteria in each group prior to starting adductor canal infusion will be documented every 6 hourly. WOMAC scores will be collected from the orthopedic database pre-operatively and at three months postoperatively.

Block performance time, pain scores on movement and rest, time to first request and the frequency of analgesic consumption, site of predominant pain, total analgesic consumption every 12 hourly and time to first physiotherapy will be documented. Intraoperative sedation requirement and intraoperative hemodynamics will be obtained from the anesthetic record. Motor strength will be evaluated with a dynamometer for maximum voluntary isometric contraction (MVIC) at 6 hours after the initial block, at 1800 PM on the day of surgery and thereafter at 0800 AM and 1600 PM for the next 72 hours. Time from the block performance/ end of infiltration to the first rescue analgesia will be determined as the total block duration. The time from the arrival in PACU to the attainment of discharge criteria will be determined as the time to readiness for discharge. Patient satisfaction will be documented on a visual analogue scale where 0 is totally dissatisfied and 100 is totally satisfied. Adverse events such as local anesthetic toxicity, symptomatic bradycardia (HR≤ 40), Significant hypotension (< 90mmHg systolic), neurological deficits, respiratory insufficiency will be prospectively collected. The failure rate and the number of attempts will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of 18-85 years of age, scheduled to undergo elective primary total knee arthroplasty.
2. ASA Class I, II, III
3. Good contralateral leg strength

Exclusion Criteria:

1. ASA physical status 4 or above
2. Patients who will need hospitalization due to reason other than the planned surgery.
3. Psychiatric illnesses.
4. Revision knee surgery
5. Narcotic dependency
6. Extraneous sources of chronic pain
7. Inability to provide informed consent.
8. Allergy to any of the drugs used in the study.
9. Contraindications to blocks and multimodal analgesia
10. Wheel chair bound

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 24 postoperative hour
  To note the duration of analgesia in the three different arms

SECONDARY OUTCOMES:
pain scores on movement | every 4 hours up to 24 hours
pain scores at rest | every 4 hours up to 24 hours
discharge criteria | 6 and 18 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Sugantha Ganapathy, FRCPC, Principal Investigator — LHSC, UWO, Canada
Locations (1):
- University Hospital, London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Fowler SJ, Christelis N. High volume local infiltration analgesia compared to peripheral nerve block for hip and knee arthroplasty-what is the evidence? Anaesth Intensive Care. 2013 Jul;41(4):458-62. doi: 10.1177/0310057X1304100404. PMID 23808503
- [Background] Abdallah FW, Brull R. Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth. 2013 Jun;110(6):915-25. doi: 10.1093/bja/aet066. Epub 2013 Apr 15. PMID 23587874